CLINICAL TRIAL: NCT00044005
Title: A Randomized, Open-Label, Dose-Blinded, Multicenter, 6-Month Study of Safety and Tolerability of 3 Dose Levels of SM-13496 (Lurasidone) in Patients With Schizophrenia
Brief Title: Safety and Tolerability Study of Drug to Treat Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1050174
Record Dates: First submitted 2002-08-16; First posted 2002-08-20 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Latuda; Lurasidone
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lurasidone 20 mg (Experimental): Lurasidone 20 mg oral tablet
  Interventions: Drug: Lurasidone 20 mg
- Lurasidione 40 mg (Experimental): Lurasidone 40 mg oral tablet
  Interventions: Drug: Lurasidone 40 mg
- Lurasidone 80mg (Experimental): Lurasidone 80mg oral tablet
  Interventions: Drug: Lurasidone 80mg

INTERVENTIONS:
Drug: Lurasidone 20 mg — Lurasidone 20mg oral tablet taken once daily for 6-months
  Arms: Lurasidone 20 mg
Drug: Lurasidone 40 mg — Lurasidone 40mg oral tablets taken once daily
  Arms: Lurasidione 40 mg
Drug: Lurasidone 80mg — Lurasidone 80mg oral tablet taken once daily
  Arms: Lurasidone 80mg

SUMMARY:
The purpose of this study is to evaluate the long-term safety of SM-13496 in patients with schizophrenia.

ELIGIBILITY:
Inclusion criteria:

* Successful completion of participation in protocol #D1050049

Exclusion criteria:

* Substance abuse
* Prolactin level of ≥200ng/mL at baseline
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2002-09; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (26):
- United States (26):
  - Birmingham Psychiatry Pharmaceutical, Birmingham, Alabama
  - Institute for Psychopharmacology Research, Cerritos, California
  - CNS Network, Garden Grove, California
  - California Clinical Trials Medical Group, Glendale, California
  - Optimum Health Services, La Mesa, California
  - University of California, Irvine, Orange, California
  - California Neuropsychopharmacology Clinical Research Institute, San Diego, California
  - Psychiatric Institute of Washington, Washington D.C., District of Columbia
  - Comprehensive Neuroscience. Inc., Melbourne, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - University of South Florida, Tampa, Florida
  - Coordinated Research of Florida, Inc, Winter Park, Florida
  - Hawaii Research Center, Honolulu, Hawaii
  - Alexian Brothers Behavioral Health Hospital, Hoffman Estates, Illinois
  - American Medical Research, Oak Brook, Illinois
  - Lake Mead Hospital, North Las Vegas, Nevada
  - Comprehensive Clinical Research, CNS, Clementon, New Jersey
  - ClinSearch, Inc., Kenilworth, New Jersey
  - Quantum Clinical Services Group, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Community Clinical Research, Austin, Texas
  - FutureSearch Trials, Austin, Texas
  - Claghorn Lesem Research Clinic, Inc., Bellaire, Texas
  - St. Paul Medical Center, Dallas, Texas
  - CNS, Inc., Falls Church, Virginia
  - Medstream, Inc., Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Lurasidone 20 mg: Lurasdione 20 mg oral tablets
- Lurasidone 40 mg: Lurasidone 40 mg oral tablets
- Lurasidone 80mg: Lurasidone 80mg oral tablets
Period: Overall Study
Arm/Group | Lurasidone 20 mg | Lurasidone 40 mg | Lurasidone 80mg
Started | 32 | 33 | 33
Completed | 13 | 19 | 11
Not Completed | 19 | 14 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lurasidone 20 mg | Lurasidone 40 mg | Lurasidone 80mg | Total
Number analyzed (Participants) | 32 | 33 | 33 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (7.8) | 42.2 (12.4) | 40.8 (10.7) | 41.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 5 | 28
  Male | 21 | 21 | 28 | 70
Region of Enrollment [Number; unit: participants]
  United States | 32 | 33 | 33 | 98

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: The primary objective of this 6-month open-label study was to evaluate the safety of 3 doses of lurasidone.
Time Frame: 6-months
Population: No formal hypothesis testing was performed. However,descriptive statistics were provided and data summarized. Safety analyses were conducted on the safety population, that included all subjects who had received at least 1 dose of open-label study medication.
Measure: Number; unit: participants
Arm/Group | Lurasidone 20 mg | Lurasidone 40 mg | Lurasidone 80mg
Number analyzed (Participants) | 32 | 33 | 33
participants | 19 (7.8) | 22 (12.4) | 18 (10.7)

ADVERSE EVENTS:
Arm/Group | Lurasidone 20 mg | Lurasidone 40 mg | Lurasidone 80mg
Serious Adverse Events (participants affected / at risk) | 3/32 | 6/33 | 3/33
Other Adverse Events (participants affected / at risk) | 19/32 | 22/33 | 18/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Lurasidone 20 mg (N=32) | Lurasidone 40 mg (N=33) | Lurasidone 80mg (N=33)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 6/6 (6) | 3/3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1)
Suicidal Behavior (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Endotracheal Intubation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lurasidone 20 mg (N=32) | Lurasidone 40 mg (N=33) | Lurasidone 80mg (N=33)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Eye Pain (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Salivary Hypersecretion (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 3 (3) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3) | 2 (2) | 3 (3)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Oedema Peripheral (General disorders) | 0 (0) | 2 (2) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (4) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 3 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 2 (2) | 1 (1) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Weight Increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Akathisia (Nervous system disorders) | 2 (2) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 6 (6) | 1 (1)
Dyskinesia (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 5 (5) | 5 (5)
Sedation (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 1 (1)
Depressed Mood (Psychiatric disorders) | 2 (2) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No